CLINICAL TRIAL: NCT02627716
Title: Effectiveness of a Joint Crisis Plan (SOS Plan) in Preventing Relapses in Patients Diagnosed With Schizophrenia and Schizoaffective Disorder
Brief Title: Joint Crisis Plan Effectiveness in Preventing Relapses in Schizophrenia and Schizoaffective Disorder
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014_04; 2014-A00911-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-07-06; First posted 2015-12-11 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2020-09

CONDITIONS: Schizophrenia
Keywords: Psychiatric advanced directives; Joint crisis plan; Schizophrenia; Primary care
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOS Intervention Group (Experimental): Subjects benefit from the SOS Plan in addition to the usual follow-ups
  Interventions: Procedure: SOS Plan
- Control Group (No Intervention): Subjects receive no additional intervention (tracking the continuation of psychiatric care according to the standard care terms)

INTERVENTIONS:
Procedure: SOS Plan — It is a customised procedure that involves a meeting (crisis planning meeting) with the patient, their various medical and social referrers and any other person who they may have desired to invite.
  The booklet outlines four avenues to consider:
  * Contact details / contact person
  * Treatment and current follow-ups
  * Medical care in the event of a crisis
  * Practical aid in the event of a crisis
  Updating the SOS Plan every 6 months in the absence of hospitalisation or after each relapse that leads to an unscheduled psychiatric hospitalisation lasting more than two weeks.
  Other Names: Joint Crisis Plan
  Arms: SOS Intervention Group

SUMMARY:
The Joint Crisis Plan = SOS Plan is a reference to a particular form of psychiatric advance directive which involves the patient, the healthcare team, their relatives and a third party caregiver as intermediary for the project.

The main objective is to evaluate the effectiveness of the SOS Plan (JCP) in terms of the reduction in hospitalisations within 18 months of its development by comparison to the standard psychiatric care.

Thus, the investigators' proposal is that SOS Plan's are regularly reassessed every 6 months and again where there is an unplanned psychiatric readmission that lasts beyond two weeks.

Single blind multicentre randomised trial with parallel control groups.

Effectiveness study of a psychiatric care strategy.

DETAILED DESCRIPTION:
Single blind multicentre randomised trial with parallel control groups.

2 groups:

* SOS Intervention Group: benefits from the SOS Plan in addition to the usual follow-ups
* "Control" Group: receive no additional intervention (only receive the routine follow-ups)

OBJECTIVES :

* To evaluate the effectiveness of the SOS Plan (JCP) in terms of the reduction in hospitalisations within 18 months of its development by comparison to the standard psychiatric care
* To evaluate :

  1. the cumulative length of hospitalisations (in days) in the two years following the development of the SOS plan
  2. the type of hospitalisation (voluntary or compulsory)
  3. the number of hospitalisations for a given subject
  4. the number of crisis situations that may require the use of the SOS Plan
  5. the clinical condition of the patient
  6. the patient with the most responses to the SOS Plan in socio-demographic terms
  7. the patient satisfaction in using the SOS Plan
  8. the decisional autonomy during treatment
  9. the quality of the therapeutic alliance
  10. the length of the meeting to develop the SOS Plan
  11. the quality of life
  12. the medico-economic impact

EXECUTION OF PRACTICAL RESEARCH :

1. The inclusion visit will be completed apart from a period of acute psychiatric decompensation, while the patient is capable of consenting to treatment. The inclusion visit will be completed within a hospital department before the patient is finally released from hospitalisation or during an outpatient follow-up.

   This involves placing the patient on the Positive And Negative Syndrome Scale (PANSS) to ensure that the patient's clinical condition allows him to consent to treatment. A score above 95 excludes the patient.

   The investigator also outlines the study and schedules visits. The patient then signs both the information letter and informed consent.

   A urine pregnancy test will be carried out on women of childbearing age.
2. Randomisation will be performed by a member of the SOS regional-referral team.

For patients in the SOS Intervention group:

* Preparatory interview with an SOS regional referrer
* SOS Plan development meeting in the presence of the patient, the treating psychiatrist, one or more relatives, and an SOS regional referrer

For patients in the control group: tracking the continuation of psychiatric care according to the standard care terms

3 ) Follow-up visits: for the two groups: 4 visits M6, M12, M18, M24 At each visit: meeting with an independent regional SOS assessor blind to allocation.

For both of the groups:

* Assessment of the clinical condition: placement on the PANSS scale
* Number of psychiatric hospitalisations, types of hospitalisation, duration of hospitalisation since the last visit
* Satisfaction assessment (numeric scale), of the therapeutic alliance (WAI), of decision-making autonomy (API), of quality of life (SF-36)

For the SOS Intervention group:

* Updating the SOS Plan after each relapse that leads to an unscheduled psychiatric hospitalisation lasting more than two weeks.
* Updating the SOS Plan every 6 months in the absence of hospitalisation

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosed with schizophrenia or schizoaffective disorder according to criteria specified in DSM
* Psychiatric inpatient or an outpatient with a specialised framework of psychiatric follow-ups
* Patient has been hospitalised at least once in a psychiatric department within the previous 2 years
* Adults under protective measures can be included (guardianship/supervision). Consent will also be sought from the guardian or trusted person.
* Registered for social security

Exclusion Criteria:

* Refusal to participate in the study
* Unable to give his or her written consent
* Patients detained
* Pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2014-12-05 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-03-10 (Actual)

PRIMARY OUTCOMES:
incidence of the first psychiatric hospitalisation | 18 months
  the incidence of the first psychiatric hospitalisation within 18 months following inclusion

SECONDARY OUTCOMES:
cumulative time in days of psychiatric hospitalisations | 2 years
  the cumulative time, in days, of psychiatric hospitalisations in the two years following inclusion
types of psychiatric hospitalisations | 2 years
  the types of psychiatric hospitalisation: voluntary (SL) or compulsory (SDT)
number of hospitalisations | 2 years
  the number of hospitalisations for each subject
number of emergency psychiatric consultations | 2 years
  the number of emergency psychiatric consultations
clinical assessment by the PANSS scale | every 6 months during 2 years
  PANSS score (intensity and qualitative aspects of the clinical situation)
patient satisfaction | every 6 months during 2 years
  score at a numeric scale of patient satisfaction
Autonomy Preference Index | every 6 months during 2 years
  decision making-autonomy assessment
Working Alliance Inventory | every 6 months during 2 years
  the working alliance assessment
length of the meeting to develop the SOS Plan | every 6 months during 2 years
  the length of the meeting to develop the SOS Plan in minutes
SF-36 quality of life | every 6 months during 2 years
  quality of life assessment by the SF-36
medical cost | every 6 months during 2 years
  numbers of hospitalisations, of consultations, drugs consummation

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Vaiva, Principal Investigator — University Hospiltal Lille
Locations (4):
- France (4):
  - University Hospital, Brest, Brest
  - University Hospital, Caen, Caen
  - University Hosiptal, Lille, Lille
  - Sainte-Anne Hospital, Paris, Paris